CLINICAL TRIAL: NCT04463836
Title: P-CLESA: Phenotyping Circulating and Lung Resident Eosinophils in Severe Asthma
Brief Title: Phenotyping Circulating and Lung Resident Eosinophils in Severe Asthma (P-CLESA)
Acronym: P-CLESA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: P82746
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Title: Phenotyping circulating and lung resident eosinophils in severe asthma (3 years).

Background: Asthma is a long-term condition that affects the airways. When a person with asthma comes into contact with something that irritates their sensitive airways, the lungs respond with contracting the muscles around the airway tubes, an inflammation process and mucus production. The airway will become narrower and inflamed making it hard to breathe and results in symptoms such as wheezing and coughing. The treatment of asthma consists of using inhalers that work to widen the airway to relief these symptoms. Often severe asthmatics have difficulty in controlling their disease, despite good medical care and taking asthma medicines. At the moment there is no cure for asthma. A new medicine called Mepolizumab (anti-Interleukin(IL)-5 therapy) has now shown to improve the symptoms of asthma particularly patients with severe asthma in whom the normal medicines prescribed for asthma are not highly effective in controlling their disease. You have been chosen receive this new medicine as we believe it will improve the control of your disease. The aim for this study is to understand the effect of Mepolizumab on a particular type of cell, called an eosinophil, which in present lungs and blood of all people but is increased in asthma patients.

Rationale: The relationship between subsets of circulating and lung resident eosinophils in severe asthma and Mepolizumab (anti-IL-5 therapy) efficacy has not been explored.

Objectives: To determine the gene expression and release of inflammatory proteins (mediator profiles) of eosinophils from the circulation and the lung, specifically blood and tissue resident, in patients with severe asthma at baseline and on Mepolizumab therapy.

Study 1: Phenotype subsets of circulating eosinophils in patients with severe asthma at one time-point Recruit: 15 biologic naïve SA and 15 SA currently on Mepo therapy. Blood eosinophils will be isolated by negative selection. Single-cell RNA-seq 10xGenomics and bulk-RNA-seq to be used to simultaneously measure gene and cell surface protein expression in the same cell to understand cellular heterogeneity in asthmatic eosinophils and identify novel targets and biomarkers for non-responsiveness Study 2: Phenotype subsets of circulating and lung eosinophils in patients with severe asthma on Mepolizumab therapy over one year.

Treat 30 appropriately characterised severe asthmatics (Eos>300/ul) with Mepolizumab Blood eosinophils will be isolated by negative selection. Single-cell RNA-seq 10xGenomics and bulk -RNA -seq to be used to understand cellular heterogeneity in asthmatic eosinophils post Mepo Therapy. Sampling at baseline, 3 and 12 months post Mepo Therapy.

Bronchoscopy performed on 30 patients, sampling endobronchial lung biopsy at baseline and 1 yr post Mepo Therapy. Single-cell RNA-seq 10xGenomics on lung resident eosinophils at baseline and 1yr post Mepolizumab therapy. Immunohistochemistry will also be performed to characterise cellular content and structure.

DETAILED DESCRIPTION:
Background: Severe asthma has been defined as "asthma which requires treatment with high dose inhaled corticosteroids (ICS) plus a second controller (and/or systemic corticosteroids) to prevent it from becoming 'uncontrolled' or which remains 'uncontrolled' despite this therapy" (1), representing a most difficult group of participants to manage. It is a heterogeneous condition and the use of mathematical approaches led to the definition of clinical subtypes (phenotypes) from cohorts in Europe, USA and Asia. With the introduction of monoclonal antibody therapies such as anti-IgE antibody (omalizumab), anti-Interleukin (IL)-5/anti-IL5Rα antibody (Mepolizumab, reslizumab and benralizumab) and anti-IL4Rα (dupilumab), personalised medicine has been initiated as these therapies are effective in patients with allergic and/or in asthma patients with increased numbers of a particular type inflammatory cell called an eosinophil (eosinophilic asthma), respectively. Introduction of these targeted therapies has helped a proportion of participants with severe asthma particularly those with eosinophilic severe asthma, but further progress will come with a better understanding of all the driving pathways underlying these phenotypes.

The biology and function of the Eosinophil Eosinophils are characterised by the presence of specific secondary granules, in their cytoplasm, containing toxic cationic proteins(2). Research studies on eosinophil biology indicate that eosinophils function in many ways including cytokine production and the development of airway inflammation. Under physiological conditions, only small numbers of eosinophils are released from the bone marrow. However, eosinophil production is dramatically increased as a result of so-called Th2 cell responses associated with allergic diseases such as asthma (2-4). There is also evidence that eosinophils contribute to homeostatic immune processes (4, 5). This increase in eosinophil production is driven by a dedicated set of cytokines, namely IL-3, IL-5, and granulocyte macrophage-CSF (GM-CSF) (2, 4). Amongst these, the Th2-associated cytokine IL-5 is the most specific cytokine for the eosinophil lineage and is responsible for the expansion of eosinophils from committed bone marrow progenitors, their release into the blood and their survival following migration into the tissues(2, 4, 6). At the site of injury, eosinophils can release their cytotoxic granule proteins as well as preformed cytokines and lipid mediators, to exacerbation of inflammation and tissue damage, which is particularly deleterious when Th2 responses are directed against allergens (2, 4).

Recruitment of eosinophils from the circulation requires blood eosinophils to become activated, leading to their attachment to activated endothelium and movement of white blood cells from the capillaries to the tissues surrounding them (extravasation(7, 8)). Arrest of eosinophils in vessels and their extravasation into the airway wall and through the bronchial tissue and epithelium to the airway lumen are mediated by a set of proteins called integrins(7, 8). Blood eosinophils from subjects with allergy or asthma, have a greater degree of adhesion or migration compared to those from normal volunteers (9).

Pharmacodynamic biomarkers for Mepolizumab treatment response Mepolizumablizumab binds with high specificity and affinity to human IL-5(10), the key T2 cytokine responsible for regulation of blood and tissue eosinophils(11). Mepolizumab prevents IL-5 from binding to the IL-5 receptor complex expressed on the eosinophil cell surface and thus inhibits IL-5 signaling, blocking eosinophil survival and proliferation. Although the exact mechanism of action of IL-5 inhibitors is not fully elucidated, the desired goal is to neutralize the effect of activated eosinophils in blood and tissues and lung, particularly the lung for asthma in order to achieve therapeutic effect.

In asthma, an association between eosinophil overexpression and asthma severity was made in 1990(12) and subsequent studies have since repeated the view that blood, or sputum eosinophil counts can be used to characterize participants with severe eosinophilic asthma (13). In the SIRIUS trial Mepolizumab at a dose of 100 mg administered subcutaneously was shown to reduce the requirement for daily oral corticosteroids while at the same time improving asthma control, lung function, and quality of life and reduced exacerbations(14). In the MENSA trial participants treated with Mepolizumab reported significantly reduced exacerbations and an improvement in asthma control questionnaire scores(15). The Mepolizumab investigators identified blood eosinophils, rather than sputum eosinophils, as a good predictor of the clinical efficacy of Mepolizumab, providing an accessible biomarker for severe eosinophilic asthma. Moreover, secondary analysis(16) of the DREAM(17) and MENSA(15) studies identified clinical efficacy of Mepolizumab in severe asthma participants with baseline eosinophil counts of ≥150-300 cells/µl and ≥300 cells/µl.

Subsets of eosinophils in asthma In mice subsets of eosinophils have been identified(18): i) lung resident eosinophils (rEos) that are IL-5-independent cells with a ring-shaped nucleus and ii) inflammatory eosinophils (iEos), which were defined as IL-5-dependent cells with a segmented nucleus. In a murine model of asthma, Mesnil and colleagues reported that the features of lung rEos remained unchanged but rEos were co-localised with iEos in the lung and that mice lacking rEos had an increased Th2 cell response to inhaled allergens. Studies in man reported that parenchymal rEos found in non-asthmatic human lungs were phenotypically distinct from the iEos isolated from the sputa of eosinophilic asthmatic patients. These data highlight the existence of distinctive circulatory and lung resident subsets of eosinophils in man.

Eosinophils secrete many molecules involved in asthma pathology including cytotoxic granule constituents cytokines and chemokines such as, lipid mediators leukotrienes(2, 19). While the role of IL-5 is a confirmed in eosinophil activation and asthma, the comparative activities of other cytokines such as GM-CSF and IL-3, also implicated in asthma, are yet to be fully determined. Eotaxins (CCL11 and CCL24) are considered to be important chemokines involved in the recruitment of eosinophils into the airways while IL-4 and IL-3 are reported to be overexpressed in the airways of severe asthmatics(20, 21). In addition to these Th2-type cytokines, IFNs and TNFα also upregulate eosinophils and prolong their survival(22, 23). Furthermore, the receptors TSLPR, IL33R and CCR3 present on activated eosinophils were found to be elevated in severe eosinophilic asthma (24) Thus, an investigation of cytokine stimulation of subsets of eosinophils, the possible crosstalk between stimulated eosinophils and the resulting differential mediator release and protein expression will likely provide a better understanding of the underlying pathophysiological signaling pathways involved in severe asthma.

Observational Study This will be an observational study of participants diagnosed with severe asthma being followed up and managed according to agreed UK guidelines for management of severe asthma. In this group, participants will have been treated with Mepolizumab according to the blood eosinophil count. These participants will be recruited and phenotyped according to eosinophilic molecular phenotype by analysis of blood and lung transcriptomics and proteomics. Participants will be evaluated at 0, 3 and 12 months. Incidental clinical finding will be forwarded to the clinical team and GP, as warranted.

Study Rationale The relationship between subsets of circulating and lung resident eosinophils in severe asthma and anti-IL-5 therapy efficacy has not been explored.

Objectives To determine the transcriptomic and mediator profiles of eosinophils from the circulation and the airway, specifically blood and tissue resident, in participants with severe asthma at baseline and on Mepolizumablizumab therapy.

Study Model Unbiased study to identify all subsets of circulating and lung resident eosinophils in biologic naïve participants with severe asthma at baseline and at time-points post treatment with Mepolizumab (anti-IL-5 Rx). Severe asthma participants (Eos>300/ul) will be recruited from the Severe Asthma clinic at the Royal Brompton Hospital, and, as much as feasible, participants will not be on OCS therapy.

Primary Objectives (i) Phenotype subsets of circulating eosinophils from participants with severe asthma at one time-point (ii) Phenotype subsets of circulating and lung eosinophils from participants with severe asthma on Mepolizumab therapy over one year.

Study 1: Phenotype subsets of circulating eosinophils in participants with severe asthma at one time-point

Recruit: 15 biologic naïve SA not on maintenance OCS and 15 SA currently on Mepolizumab therapy with good clinical response.

Blood samples (90ml) will be taken from these participants. Blood eosinophils will be isolated from these samples which will then be subtyped (phenotype) by simultaneously measuring gene and cell surface protein expression in the same cell. Blood eosinophils will also be cell-cultured in the laboratory and stimulated with a variety of cytokines and chemokines the release of inflammatory mediators determined. Together, this will increase our understanding of the cellular heterogeneity in asthmatic eosinophils and identify the difference between peripheral blood eosinophil populations in untreated and Mepolizumablizumab treated participants .

Study 2: Phenotype subsets of circulating and lung eosinophils from participants with severe asthma on Mepolizumab therapy over one year.

Recruit 36 severe asthma participants appropriately characterised severe asthmatics (Eos>300/ul), not on OCS maintenance therapy, to achieve paired biopsy samples from 30 participants

Blood samples will be taken at baseline, 3 and 12 months post-Mepolizumab Therapy. Blood eosinophils will then be isolated and phenotyped by simultaneously measuring gene and cell surface protein expression in the same cell. Blood eosinophils will also be cell-cultured in the laboratory and stimulated with a variety of cytokines and chemokines the release of inflammatory mediators determined. Together, this will increase our understanding of cellular heterogeneity in asthmatic eosinophils post Mepolizumab Therapy.

Bronchoscopy will be performed on 36 participants, sampling endobronchial lung biopsy at baseline and 1 yr post Mepolizumab Therapy; the second procedure will be performed within 2 weeks of the last Mepolizumab injection. Single-cell RNA-seq 10xGenomics and bulk -RNA -seq will be performed, using the optimized protocol of the Gronigen group, on lung tissue eosinophils through enzymatic disassociation of lung tissue (at 4oC) at baseline and 1yr post Mepolizumab therapy. Immunohistochemistry (IHC) will also be performed to characterise cellular content and structure. Four biopsies will be reserved for RNA-seq and two for IHC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged between 18 years and 70 years.
* Give written informed consent prior to participation in the study including all of its procedures.
* Comply with study protocol requirements
* Able to read, comprehend, and write at a sufficient level to complete study related materials.
* Able to complete the study and all measurements.
* All participants have been through a severe asthma protocol that have ascertained the diagnosis of severe asthma, maximised treatments and ensured adherence to therapy.
* Stable asthma therapy for at least a month before screening
* On <10 mg maintenance OCS therapy

Exclusion criteria:

Subjects will not be eligible if any of the following apply: -

* As a result of medical interview, physical examination or screening investigation the investigators consider the subject unfit either because of risk to the subject due to the study or the influence this may have on the study results.
* A history of recreational drug use or allergy which in the opinion of the investigators contra-indicates their participation.
* Participation within 3 months in any a trial testing a new molecular entity or drug.
* Those, in the opinion of the investigator, who may prove non-compliant with study procedures.
* Within 4 weeks of screening visit been hospitalized or required high dose oral corticosteroid (>30 mg prednisolone per day) therapy, asthma not been stable.
* Participants who have had prior treatment with bronchial thermoplasty, defined as completion of all thermoplasty treatment sessions within 6 months of screening
* History of significant pulmonary disease other than severe asthma.
* History of pulmonary eosinophilic syndrome or hyper eosinophilic syndrome.
* History of bronchopulmonary aspergillosis

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All the participants identified as being eligible with severe asthma confirmed by a multidisciplinary team in the Royal Brompton Hospital will be invited to take part in the study. Participants referred to the severe asthma clinic will undergo a specific protocol that leads to the ultimate diagnosis of severe asthma as defined by the ERS/ATS guidelines for severe asthma (1). Participants with severe asthma will be diagnosed as persistently poor control and/or exacerbations of asthma despite high dose therapy defined as at least 1000 μg fluticasone propionate equivalent per day and a second controller. The evaluation will include an assessment of adherence to therapies.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Phenotype subsets of circulating eosinophils from participants with severe asthma at one time-point | 18 months
  Determine the transcriptomic and mediator profiles of eosinophils from the circulation, specifically blood, in participants with severe asthma on Mepolizumab therapy.
Phenotype subsets of circulating and lung eosinophils from participants with severe asthma on Mepolizumab therapy over one year. | 3 years
  Determine the transcriptomic and mediator profiles of eosinophils from the circulation and the airway, specifically blood and tissue resident, in participants with severe asthma at baseline and on Mepolizumab therapy at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj K Bhavsar, PhD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton & Harefield NHS Trust,, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Transcriptomic and mediator profiles, in terms pseudonymised samples, will be sent to the Netherlands
Supporting Information: Study Protocol
Time Frame: 18 months - 4 years from start of study

REFERENCES:
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Background] Rothenberg ME, Hogan SP. The eosinophil. Annu Rev Immunol. 2006;24:147-74. doi: 10.1146/annurev.immunol.24.021605.090720. PMID 16551246
- [Background] Travers J, Rothenberg ME. Eosinophils in mucosal immune responses. Mucosal Immunol. 2015 May;8(3):464-75. doi: 10.1038/mi.2015.2. Epub 2015 Mar 25. PMID 25807184
- [Background] Rosenberg HF, Dyer KD, Foster PS. Eosinophils: changing perspectives in health and disease. Nat Rev Immunol. 2013 Jan;13(1):9-22. doi: 10.1038/nri3341. Epub 2012 Nov 16. PMID 23154224
- [Background] Chu VT, Beller A, Rausch S, Strandmark J, Zanker M, Arbach O, Kruglov A, Berek C. Eosinophils promote generation and maintenance of immunoglobulin-A-expressing plasma cells and contribute to gut immune homeostasis. Immunity. 2014 Apr 17;40(4):582-93. doi: 10.1016/j.immuni.2014.02.014. PMID 24745334
- [Background] Lopez AF, Sanderson CJ, Gamble JR, Campbell HD, Young IG, Vadas MA. Recombinant human interleukin 5 is a selective activator of human eosinophil function. J Exp Med. 1988 Jan 1;167(1):219-24. doi: 10.1084/jem.167.1.219. PMID 2826636
- [Background] Johansson MW, Mosher DF. Integrin activation States and eosinophil recruitment in asthma. Front Pharmacol. 2013 Apr 1;4:33. doi: 10.3389/fphar.2013.00033. eCollection 2013. PMID 23554594
- [Background] Barthel SR, Johansson MW, McNamee DM, Mosher DF. Roles of integrin activation in eosinophil function and the eosinophilic inflammation of asthma. J Leukoc Biol. 2008 Jan;83(1):1-12. doi: 10.1189/jlb.0607344. Epub 2007 Oct 10. PMID 17906117
- [Background] Hakansson L, Heinrich C, Rak S, Venge P. Priming of eosinophil adhesion in patients with birch pollen allergy during pollen season: effect of immunotherapy. J Allergy Clin Immunol. 1997 Apr;99(4):551-62. doi: 10.1016/s0091-6749(97)70084-8. PMID 9111502
- [Background] Hart TK, Cook RM, Zia-Amirhosseini P, Minthorn E, Sellers TS, Maleeff BE, Eustis S, Schwartz LW, Tsui P, Appelbaum ER, Martin EC, Bugelski PJ, Herzyk DJ. Preclinical efficacy and safety of mepolizumab (SB-240563), a humanized monoclonal antibody to IL-5, in cynomolgus monkeys. J Allergy Clin Immunol. 2001 Aug;108(2):250-7. doi: 10.1067/mai.2001.116576. PMID 11496242
- [Background] Chung KF. Targeting the interleukin pathway in the treatment of asthma. Lancet. 2015 Sep 12;386(9998):1086-96. doi: 10.1016/S0140-6736(15)00157-9. PMID 26383000
- [Background] Bousquet J, Chanez P, Lacoste JY, Barneon G, Ghavanian N, Enander I, Venge P, Ahlstedt S, Simony-Lafontaine J, Godard P, et al. Eosinophilic inflammation in asthma. N Engl J Med. 1990 Oct 11;323(15):1033-9. doi: 10.1056/NEJM199010113231505. PMID 2215562
- [Background] Yancey SW, Keene ON, Albers FC, Ortega H, Bates S, Bleecker ER, Pavord I. Biomarkers for severe eosinophilic asthma. J Allergy Clin Immunol. 2017 Dec;140(6):1509-1518. doi: 10.1016/j.jaci.2017.10.005. PMID 29221581
- [Background] Bel EH, Wenzel SE, Thompson PJ, Prazma CM, Keene ON, Yancey SW, Ortega HG, Pavord ID; SIRIUS Investigators. Oral glucocorticoid-sparing effect of mepolizumab in eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1189-97. doi: 10.1056/NEJMoa1403291. Epub 2014 Sep 8. PMID 25199060
- [Background] Ortega HG, Liu MC, Pavord ID, Brusselle GG, FitzGerald JM, Chetta A, Humbert M, Katz LE, Keene ON, Yancey SW, Chanez P; MENSA Investigators. Mepolizumab treatment in patients with severe eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1198-207. doi: 10.1056/NEJMoa1403290. Epub 2014 Sep 8. PMID 25199059
- [Background] Ortega HG, Yancey SW, Mayer B, Gunsoy NB, Keene ON, Bleecker ER, Brightling CE, Pavord ID. Severe eosinophilic asthma treated with mepolizumab stratified by baseline eosinophil thresholds: a secondary analysis of the DREAM and MENSA studies. Lancet Respir Med. 2016 Jul;4(7):549-556. doi: 10.1016/S2213-2600(16)30031-5. Epub 2016 May 10. PMID 27177493
- [Background] Pavord ID, Korn S, Howarth P, Bleecker ER, Buhl R, Keene ON, Ortega H, Chanez P. Mepolizumab for severe eosinophilic asthma (DREAM): a multicentre, double-blind, placebo-controlled trial. Lancet. 2012 Aug 18;380(9842):651-9. doi: 10.1016/S0140-6736(12)60988-X. PMID 22901886
- [Background] Mesnil C, Raulier S, Paulissen G, Xiao X, Birrell MA, Pirottin D, Janss T, Starkl P, Ramery E, Henket M, Schleich FN, Radermecker M, Thielemans K, Gillet L, Thiry M, Belvisi MG, Louis R, Desmet C, Marichal T, Bureau F. Lung-resident eosinophils represent a distinct regulatory eosinophil subset. J Clin Invest. 2016 Sep 1;126(9):3279-95. doi: 10.1172/JCI85664. Epub 2016 Aug 22. PMID 27548519
- [Background] Hogan SP, Rosenberg HF, Moqbel R, Phipps S, Foster PS, Lacy P, Kay AB, Rothenberg ME. Eosinophils: biological properties and role in health and disease. Clin Exp Allergy. 2008 May;38(5):709-50. doi: 10.1111/j.1365-2222.2008.02958.x. Epub 2008 Apr 1. PMID 18384431
- [Background] Wenzel S, Wilbraham D, Fuller R, Getz EB, Longphre M. Effect of an interleukin-4 variant on late phase asthmatic response to allergen challenge in asthmatic patients: results of two phase 2a studies. Lancet. 2007 Oct 20;370(9596):1422-31. doi: 10.1016/S0140-6736(07)61600-6. PMID 17950857
- [Background] Wenzel S, Ford L, Pearlman D, Spector S, Sher L, Skobieranda F, Wang L, Kirkesseli S, Rocklin R, Bock B, Hamilton J, Ming JE, Radin A, Stahl N, Yancopoulos GD, Graham N, Pirozzi G. Dupilumab in persistent asthma with elevated eosinophil levels. N Engl J Med. 2013 Jun 27;368(26):2455-66. doi: 10.1056/NEJMoa1304048. Epub 2013 May 21. PMID 23688323
- [Background] Kankaanranta H, Ilmarinen P, Zhang X, Adcock IM, Lahti A, Barnes PJ, Giembycz MA, Lindsay MA, Moilanen E. Tumour necrosis factor-alpha regulates human eosinophil apoptosis via ligation of TNF-receptor 1 and balance between NF-kappaB and AP-1. PLoS One. 2014 Feb 28;9(2):e90298. doi: 10.1371/journal.pone.0090298. eCollection 2014. PMID 24587316
- [Background] Letuve S, Druilhe A, Grandsaigne M, Aubier M, Pretolani M. Involvement of caspases and of mitochondria in Fas ligation-induced eosinophil apoptosis: modulation by interleukin-5 and interferon-gamma. J Leukoc Biol. 2001 Nov;70(5):767-75. PMID 11698497
- [Background] Kuo CS, Pavlidis S, Zhu J, Loza M, Baribaud F, Rowe A, Pandis I, Gibeon D, Hoda U, Sousa A, Wilson SJ, Howarth P, Shaw D, Fowler S, Dahlen B, Chanez P, Krug N, Sandstrom T, Fleming L, Corfield J, Auffray C, Djukanovic R, Sterk PJ, Guo Y, Adcock IM, Chung KF; U-BIOPRED Project Team. Contribution of airway eosinophils in airway wall remodeling in asthma: Role of MMP-10 and MET. Allergy. 2019 Jun;74(6):1102-1112. doi: 10.1111/all.13727. Epub 2019 Feb 11. PMID 30667542